CLINICAL TRIAL: NCT03558958
Title: An Exploratory, Open-label Study to Assess the Effect of P-188 NF (Carmeseal-MD) on Safety, on Respiratory and Cardiac Dysfunction and on Upper Limb Strength in Non-ambulatory Patients With Duchenne Muscular Dystrophy (DMD)
Brief Title: Safety and Efficacy of P-188 NF in DMD Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to lack of funding.
Sponsor: Phrixus Pharmaceuticals, Inc. (Industry)
Collaborators: Charley's Fund (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-004
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2021-09

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- P-188 NF (Experimental): P-188 NF, 5 mg/Kg administered subcutaneously daily for 1 year
  Interventions: Drug: P-188 NF

INTERVENTIONS:
Drug: P-188 NF — Poloxamer administered daily via sc injection at 5 mg/Kg
  Other Names: Carmeseal-MD

SUMMARY:
This is an open-label study to evaluate the safety, tolerability and efficacy of daily, subcutaneous dosing with P-188 NF (Carmeseal-MD™) in non-ambulatory boys with Duchenne Muscular Dystrophy (DMD). This study will determine if continuous treatment with Carmeseal-MD™ can maintain or improve pulmonary function, and skeletal and cardiac muscle function, compared to baseline, in boys 12-25 years of age.

DETAILED DESCRIPTION:
Based on a large number of studies conducted in pre-clinical models of muscular dystrophy and heart failure, this study is being undertaken to explore the safety and efficacy of Carmeseal-MD™ (P-188 NF) on endpoints associated with cardiovascular, pulmonary and musculoskeletal function. These preclinical studies indicate that Carmeseal-MD™ acts to stabilize fragile cell membranes thus maintaining cell function and preventing fibrosis, necrosis and apoptosis in animal models of muscular dystrophy.

This is a single arm, open label trial that is designed to provide a first evaluation of Carmeseal-MD™ in non-ambulatory patients with DMD. It assigns up to ten (10) patients to receive a fixed dose of 5 mg of P-188 NF per Kg patient body weight (adjusted individually for each patient at baseline visit) injected subcutaneously once-a-day for 52 weeks. The first 3 enrolled subjects (Group 1) will be at least 18 years of age and up to 25 years of age. Enrollment of Group 2 will begin after a review of Group 1 safety data through 28 days of dosing of Carmeseal-MD™. Group 2 will include subjects that are at least 12 years of age and up to 25 years old. Evaluations will be for Carmeseal-MD™ administered in addition to the current standard of care therapies and interventions such as corticosteroids, ACE inhibitors, ARBs, beta blockers, bronchodilator medications and airway clearance, cough assist and non-invasive ventilation devices.

The major hypothesis for the trial is that measures of function of skeletal and cardiac muscle that decline over the course of the disease will either remain stable or improve with P-188 NF treatment when a decline would be expected. To assess these possible beneficial effects, comparisons are planned between pre- and post-treatment on measures of function for the various body systems affected by DMD.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 12 - 25 years of age
* Have phenotypic evidence of DMD
* Have documentation of the presence of a deletion, duplication or point mutation in the dystrophin gene
* Willingness to receive daily subcutaneous (SC) injections of up to 3 mL
* Have LVEDV that is ≥100% of normal corrected for body mass when measured by cardiac MRI
* Have impaired respiratory function (percent predicted PEF ≤80%)
* Have ability to perform PEF within 15% of first assessment
* Have mild to moderate fibrosis of the heart as assessed by MRI
* Have left ventricular ejection fraction fractions of <50%
* Have been non-ambulatory for at least six months
* Be on corticosteroids, with a stable treatment regimen for at least six months
* Have been on a stable treatment regimen for cardiac dysfunction for at least 3 months prior to baseline (ACE inhibitors, beta blockers and/or ARBs)
* Have clinically acceptable screening values, including serum creatinine levels blood urine nitrogen, cystatin C
* Have willingness and ability to comply with scheduled visits, drug administration, drug administrative plan, study procedures, laboratory tests, and treatment restrictions
* Be likely to survive for the duration of the treatment in the investigator's opinion
* Have ability to provide written informed consent (parent/guardian consent if applicable)/assent (if <18 years of age).

Exclusion Criteria:

* Exposure to another investigational drug within 90 days prior to start of study treatment
* Have DMD-related hypoventilation for which daytime assisted ventilation is needed
* Unable to perform pulmonary function testing
* Have respiratory failure
* Unable or unwilling to undergo scan with gadolinium as contrast agent
* Unable or unwilling to undergo echocardiography
* Have severe fibrosis of the heart as assessed by MRI
* Used carnitine, creatine, glutamine, oxatomide, coenzyme Q10 or vitamin E or any herbal medicines with 30 days prior to baseline
* Have a history of major surgical procedure within 30 days prior to start of study treatment
* Have ongoing immunosuppressive therapy (other than corticosteroids)
* Are participating in a therapeutic clinical trial
* Are on any concomitant medication with a depressive or stimulating effect on respiration or the respiratory tract
* Have a diagnosis of chronic lung disease
* Chronic use of beta-2 agonists or any other bronchodilating medication (chronic use is daily intake for more than 14 days within the last 6 months)
* Have moderate or severe hepatic impairment or moderate to severe renal impairment
* Have expectation of major surgical procedure during the conduct of the study
* Have prior or ongoing medical conditions that makes it unlikely that the course of treatment or follow-up would be completed, or could impair the assessment of the treatment results
* Have ever previously received P-188 NF as a therapeutic agent

Ages: 12 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Forced vital capacity (FVC) | Baseline, Days 91, 182, 273, 364
  Change from baseline (pre-treatment) to end of treatment (52 weeks)

SECONDARY OUTCOMES:
Maximal inspiratory pressure (MIP) | Baseline, Days 91, 182, 273, 364
  Change from baseline (pre-treatment) to end of treatment (52 weeks)
Maximal expiratory pressure (MEP) | Baseline, Days 91, 182, 273, 364
  Change from baseline (pre-treatment) to end of treatment (52 weeks)
Peak cough flow (PCF) | Baseline, Days 91, 182, 273, 364
  Change from baseline (pre-treatment) to end of treatment (52 weeks)
Left ventricular end-diastolic volume (LVEDV) | Baseline, Days 91, 182, 273, 364
  Change from baseline (pre-treatment) to end of treatment (52 weeks)
Ejection Fraction (EF) | Baseline, Days 91, 182, 273, 364
  Change from baseline (pre-treatment) to end of treatment (52 weeks)
Degree of fibrosis as assessed by cardiac MRI | Baseline, Days 182, 364
  Change from baseline (pre-treatment) to end of treatment (52 weeks)
Performance of upper limb (PUL) test | Baseline, Days 91, 182, 273, 364
  Change from baseline (pre-treatment) to end of treatment (52 weeks)
Cardiac troponin I | Baseline, Days 28, 56, 91, 182, 273, 364
  Change from baseline (pre-treatment) to end of treatment (52 weeks)
Muscle creatine kinase | Baseline, Days 28, 56, 91, 182, 273, 364
  Change from baseline (pre-treatment) to end of treatment (52 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ryan, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ng R, Metzger JM, Claflin DR, Faulkner JA. Poloxamer 188 reduces the contraction-induced force decline in lumbrical muscles from mdx mice. Am J Physiol Cell Physiol. 2008 Jul;295(1):C146-50. doi: 10.1152/ajpcell.00017.2008. Epub 2008 May 21. PMID 18495816
- [Background] Ilsar, I., Wang, M., Jiang, A., Dye, K., Markham, B., Sabbah, H.N. (2010) Acute intravenous bolus injection of Poloxamer-188 improves left ventricular function in dogs with heart failure J. Am. Col. Cardiol. 55 (Suppl. 1): A16.E146.
- [Background] Townsend D, Turner I, Yasuda S, Martindale J, Davis J, Shillingford M, Kornegay JN, Metzger JM. Chronic administration of membrane sealant prevents severe cardiac injury and ventricular dilatation in dystrophic dogs. J Clin Invest. 2010 Apr;120(4):1140-50. doi: 10.1172/JCI41329. Epub 2010 Mar 15. PMID 20234088
- [Background] Houang EM, Haman KJ, Filareto A, Perlingeiro RC, Bates FS, Lowe DA, Metzger JM. Membrane-stabilizing copolymers confer marked protection to dystrophic skeletal muscle in vivo. Mol Ther Methods Clin Dev. 2015 Nov 11;2:15042. doi: 10.1038/mtm.2015.42. eCollection 2015. PMID 26623440
- [Background] Lin B, Li Y, Han L, Kaplan AD, Ao Y, Kalra S, Bett GC, Rasmusson RL, Denning C, Yang L. Modeling and study of the mechanism of dilated cardiomyopathy using induced pluripotent stem cells derived from individuals with Duchenne muscular dystrophy. Dis Model Mech. 2015 May;8(5):457-66. doi: 10.1242/dmm.019505. Epub 2015 Mar 19. PMID 25791035
- [Background] Plant DR, Ryall JG, Lynch GS. Contraction-mediated damage in mdx dystrophic mouse tibialis anterior muscles is not affected by the membrane sealant poloxamer Proc. Australia Physiological Society. 2005; 36: 133P
- [Background] Ryall JG, van der Poel C, Schertzer JD, Plant DR, Lynch GS, The membrane sealant poloxamer reduces membrane permeability in tibialis anterior muscles from dystrophic mdx mice. The FASEB Journal. 2007;21: 769.28.